CLINICAL TRIAL: NCT02532179
Title: A Biomarker-Based Pilot Study of Mouse Subcutaneous Immunotherapy in Mouse Sensitive Adults With Asthma and/or Perennial Allergic Rhinitis (ICAC-26)
Brief Title: Subcutaneous Immunotherapy for Mouse in Adults
Acronym: SCITMO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Inner-City Asthma Consortium (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ICAC-26
Record Dates: First submitted 2015-08-21; First posted 2015-08-25 (Estimated); Results first posted 2017-11-28 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Asthma; Perennial Allergic Rhinitis
Keywords: subcutaneous immunotherapy (SCIT); glycerinated mouse allergenic extract; mouse specific IgE; mouse specific IgG and IgG4; mouse prick skin test wheal
MeSH Terms: conditions — Asthma; Rhinitis, Allergic, Perennial | interventions — Urea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mouse Allergenic Extract (Experimental): Participants will receive escalating doses of glycerinated mouse allergenic extract administered via the subcutaneous route up to a Maximum Study Dose (MSD) of 0.4 mL of extract at a concentration of 1:10 wt/vol.
  Interventions: Biological: Mouse Allergenic Extract

INTERVENTIONS:
Biological: Mouse Allergenic Extract — Subjects will receive escalating doses of glycerinated mouse allergenic extract administered subcutaneously up to a maximum study dose (MSD) of 0.4 mL of extract at a concentration of 1:10 wt/vol., per protocol.
  Other Names: mouse epithelial extract; allergenic extract of Mus musculus

SUMMARY:
This is an open label trial of mouse allergenic extract administered by subcutaneous injection in adults with asthma and mouse sensitivity. The study is designed to evaluate:

* the safety of this therapy when given by injection
* biomarkers of the immune response and
* whether the therapy would be effective in treating allergic asthma.

DETAILED DESCRIPTION:
The primary objective of the study is to assess if treatment with mouse subcutaneous immunotherapy (SCIT), using the per protocol allergenic extract doses, is safe. This will be done by determining the rate of related adverse events and serious adverse events in the course of treatment.

Secondary objectives include:

* determination of whether a 24 week treatment with mouse SCIT, using the per protocol allergenic extract doses, will induce a 3-fold increase in mouse-specific serum immunoglobulin E (IgE)
* determination of whether a 24 week treatment with mouse SCIT, using the per protocol allergenic extract doses, will induce changes in the serum levels of mouse-specific immunoglobulin G (IgG) and immunoglobulin subclass 4 (IgG4).

ELIGIBILITY:
INCLUSION CRITERIA

Participants who meet any of the following criteria are not eligible for enrollment but may be reassessed. Participants are ineligible if they:

* Are pregnant or lactating. Females must be abstinent or use a medically acceptable birth control method throughout the study (e.g. oral, subcutaneous, mechanical, or surgical contraception);
* Cannot perform spirometry at Screening;
* Have an asthma severity classification at Recruitment of severe persistent, using the NAEPP classification, as evidenced by at least one of the following:

  * Requires a dose of greater than 500 mcg of fluticasone per day or the equivalent of another inhaled corticosteroid;
  * Have received more than 2 courses of oral or parenteral corticosteroids within the last 12 months;
  * Have been treated with depot steroids within the last 12 months;
  * Have been hospitalized for asthma within the 6 months prior to recruitment;
  * Have had a life-threatening asthma exacerbation that required intubation, mechanical ventilation, or that resulted in a hypoxic seizure within 2 years prior to recruitment.
* Do not have access to a phone (needed for scheduling appointments);
* Have received allergen immunotherapy (SLIT or SCIT) in the last 12 months prior to recruitment or who plan to initiate or resume allergen immunotherapy during the study;
* Have previously been treated with anti-IgE therapy within 1 year of recruitment;
* Have received an investigational drug in the 30 days prior to recruitment or who plan to use an investigational drug during the study;
* Refuses to sign the Epinephrine Auto-injector Training Form.

EXCLUSION CRITERIA

Participants who meet any of the following criteria are not eligible for enrollment and may not be reassessed. Participants are ineligible if they:

* Do not primarily speak English;
* Plan to move from the area during the study period;
* Have a history of idiopathic anaphylaxis or anaphylaxis grade 2 or higher as defined per protocol;
* Have unstable angina, significant arrhythmia, uncontrolled hypertension, history of autoimmune disease, or other chronic or immunological diseases that in the opinion of the investigator might interfere with the evaluation of the investigational agent or pose additional risk to the participant;
* Are using tricyclic antidepressants or beta-adrenergic blocker drugs (both oral and topical);
* Have not received the seasonal Flu (Influenza) Vaccine if enrolling December through March.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wood, M.D., Study Chair — Johns Hopkins Children's Center: Department of Allergy & Immunology
Locations (4):
- United States (4):
  - Children's National Health System, Washington D.C., District of Columbia
  - Ann and Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins Children's Center: Department of Allergy & Immunology, Baltimore, Maryland
  - Henry Ford Health System: Division of Allergy and Immunology, Detroit, Michigan

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: History, project and sites of the Inner-city Asthma Consortium (ICAC) — https://www.niaid.nih.gov/clinical-trials/inner-city-asthma-consortium
- See also: Information: National Asthma Education and Prevention Program (NAEPP) — http://www.nhlbi.nih.gov/about/org/naepp

RESULTS

PARTICIPANT FLOW:
Groups:
- Mouse Allergenic Extract: Participants received escalating doses of glycerinated mouse allergenic extract administered via the subcutaneous route. The first injection contained 0.05 mL of 1:10,000 concentration of 1:20 weight per volume (w/v) glycerinated mouse allergenic extract. Administration of additional dosages were given at study clinician's discretion, up to a Maximum Study Dose (MSD) of 0.4 mL of extract at a concentration of 1:10 w/v, for the first 11 weeks of the 24-week treatment with two injections per week, separated by at least 2 days. Dose escalation continued until maximum study dose was achieved in a maximum of 18 weeks. For the remaining time of the 24-week treatment, participants received one injection of investigational agent every 2 weeks and were asked to report any symptoms possibly related to the investigation agent to the study sites.
Period: Overall Study
Arm/Group | Mouse Allergenic Extract
Started | 12
Completed | 9
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Pregnancy | 1
Not completed — Subject received depot steroid injection | 1

BASELINE CHARACTERISTICS:
Arm/Group | Mouse Allergenic Extract
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (7.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 2
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Mouse-Specific Serum Immunoglobulin E (IgE) Levels [Geometric Least Squares Mean (Standard Deviation); unit: kU/L] — Serum Immunoglobulin E (IgE) is an antibody produced by the immune system. If a participant has an allergy, the immune system will respond to that particular allergen by producing antibodies called IgE. These antibodies travel to cells that release chemicals, which cause allergic reactions. We collect mouse-specific serum IgE at baseline and compare with post-baseline IgE in order to determine immune modulation over time. The higher the IgE present in the serum sample, the more likely there is to be a presence of a clinical allergy to the mouse allergen.
  kU/L | 2.34 (0.45)
Mouse-Specific Serum Immunoglobulin G (IgG) Levels [Geometric Least Squares Mean (Standard Deviation); unit: kU/L] — Serum Immunoglobulin G (IgG) is an antibody produced by the immune system. If a participant has bacterial or viral infections, the immune system will respond to that particular infection by producing antibodies called IgG. We collect mouse-specific serum IgG at baseline and compare with post-baseline IgG in order to determine immune modulation over time. The higher the IgG present in the serum sample, the more likely there is to be a presence of a clinical allergy to the mouse allergen.
  kU/L | 1.23 (0.20)
Mouse-Specific Serum Immunoglobulin G4 (IgG4) Levels [Geometric Least Squares Mean (Standard Deviation); unit: kU/L] — Serum Immunoglobulin G4 (IgG4) is a certain subtype of antibody produced by the immune system. If a participant has bacterial or viral infections, the immune system will respond to that particular infection by producing antibodies called IgG4. We collect mouse-specific serum IgG4 at baseline and compare with post-baseline IgG4 in order to determine immune modulation over time. The higher the IgG4 present in the serum sample, the more likely there is to be a presence of a clinical allergy to the mouse allergen.
  kU/L | 0.08 (0.35)

OUTCOME MEASURES:

1. Primary Outcome: Number of Reported Adverse Events (AEs)
Description: Frequency of any AEs tabulated by preferred event term.
Time Frame: Baseline (Pre-Treatment) through 24 Weeks of Treatment
Population: Intent-to-treat
Measure: Number; unit: Events
Arm/Group | Mouse Allergenic Extract
Number analyzed (Participants) | 12
Events
  Total adverse events | 9
  Abdominal pain | 1
  Vomiting | 1
  Injection site swelling | 2
  Peak expiratory flow rate decreased | 2
  Pruritus generalized | 1
  Skin lesion | 1
  Flushing | 1

2. Primary Outcome: Number of Reported Serious Adverse Events (SAEs)
Description: Frequency of any Serious Adverse Events (SAEs) throughout the duration of study participation.
Time Frame: Baseline (Pre-Treatment) through 24 Weeks of Treatment
Population: Intent-to-treat
Measure: Number; unit: Number of SAEs
Arm/Group | Mouse Allergenic Extract
Number analyzed (Participants) | 12
Number of SAEs | 0

3. Secondary Outcome: Change in Mouse-Specific IgE Antibodies
Description: Serum Immunoglobulin E (IgE) is an antibody produced by the immune system. If a participant has an allergy, the immune system will respond to that particular allergen by producing IgE antibodies. These antibodies travel to cells that release chemicals, causing allergic reactions.
  This endpoint/outcome is the ratio of geometric means for baseline mouse-specific serum IgE versus post-baseline mouse-specific serum IgE. The numerator is the geometric mean post-baseline IgE and the denominator is baseline IgE. A ratio of greater than 1 would indicate an increase in IgE throughout the course of the study.
Time Frame: Baseline (Pre-Treatment) through Week 24
Population: Intent-to-treat
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Mouse Allergenic Extract
Number analyzed (Participants) | 12
Ratio | 3 [2.09 to 4.29]
Statistical Analysis 1: Comparison: Mouse Allergenic Extract; Test type: Superiority; p < 0.001, Mixed Models Analysis — Null hypothesis: there is no difference in immune modulation over time; Mean Ratio = 3, 95% CI 2-sided [2.09 to 4.29]

4. Secondary Outcome: Change in Mouse-Specific IgG Antibodies
Description: Serum Immunoglobulin G (IgG) is an antibody produced by the immune system. If a participant has bacterial or viral infections, the immune system will respond to that particular infection by producing IgG antibodies.
  This endpoint/outcome is the ratio of geometric means for baseline mouse-specific serum IgG versus post-baseline mouse-specific serum IgG. The numerator is the geometric mean post-baseline IgG and, the denominator is the baseline IgG. A ratio of greater than 1 would indicate an increase in IgG throughout the course of the study.
Time Frame: Baseline (Pre-Treatment) to Week 24
Population: Intent-to-treat
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Mouse Allergenic Extract
Number analyzed (Participants) | 12
Ratio | 3.82 [2.77 to 5.25]
Statistical Analysis 1: Comparison: Mouse Allergenic Extract; Test type: Superiority; p < 0.001, Mixed Models Analysis — Null hypothesis: there is no difference in immune modulation over time; Mean Ratio = 3.82, 95% CI 2-sided [2.77 to 5.25]

5. Secondary Outcome: Change in Mouse-Specific IgG4 Antibodies
Description: Serum Immunoglobulin G4 (IgG4) is a subtype of antibody produced by the immune system. If a participant has bacterial or viral infections, the immune system will respond to that particular infection by producing IgG4 antibodies.
  This endpoint/outcome is the ratio of geometric means for baseline mouse-specific serum IgG4 versus post-baseline mouse-specific serum IgG4. The numerator is the geometric mean post-baseline IgG4 and, the denominator is the baseline IgG4. A ratio of greater than 1 would indicate an increase in IgG4 antibodies throughout the course of the study.
Time Frame: Baseline (Pre-Treatment) to Week 24
Population: Intent-to-treat
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Mouse Allergenic Extract
Number analyzed (Participants) | 12
Ratio | 6.55 [3.87 to 11.06]
Statistical Analysis 1: Comparison: Mouse Allergenic Extract; Test type: Superiority; p < 0.001, Mixed Models Analysis — Null hypothesis: there is no difference in immune modulation over time; Mean Ratio = 6.55, 95% CI 2-sided [3.87 to 11.06]

6. Secondary Outcome: Change in In-vitro Mouse Antigen Binding to B-cells
Description: The plan was to analyze serum from cockroach subcutaneous immunotherapy (SCIT)-treated participants to determine if treatment inhibits in-vitro mouse antigen binding to B-cells after 6-months of treatment with mouse SCIT, using the per protocol allergenic extract doses. However, the Sponsor cancelled pursuit of mouse immunotherapy within its program at this time due to assay development complexities and cost; thus, there are no analyses/results for this endpoint/outcome.
Time Frame: Baseline (Pre-Treatment) to Week 24
Population: No analysis conducted: Sponsor's decision to not pursue assay development in this study.
Arm/Group | Mouse Allergenic Extract
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Enrollment through end of study (up to 24 weeks)
Groups:
- Mouse Allergenic Extract: Participants received escalating doses of glycerinated mouse allergenic extract administered via the subcutaneous route. The first injection contained 0.05 mL of 1:10,000 concentration of 1:20 w/v glycerinated mouse allergenic extract, with proceeding administration of additional dosage at study clinician's discretion, for up to a Maximum Study Dose (MSD) of 0.4 mL of extract at a concentration of 1:10 wt/vol for the first 11 weeks of the 24-week treatment with two injections per week, separated by at least 2 days. Dose escalation would continue until maximum study dose is achieved in a maximum of 18 weeks. For the remaining time of the 24-week treatment, participants would receive one injection of investigational agent every 2 weeks and were asked to report any symptoms possibly related to the investigation agent to the study sites.
Arm/Group | Mouse Allergenic Extract
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 6/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mouse Allergenic Extract (N=12)
Injection site swelling (General disorders) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Peak expiratory flow rate decreased (Investigations) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT02532179/Prot_SAP_000.pdf